CLINICAL TRIAL: NCT07249840
Title: Pilot Study of Ropeginterferon for Patients With JAK2 V617F Clonal Hematopoiesis and High-Risk Features
Brief Title: Ropeginterferon for High Risk JAK2 Clonal Hematopoiesis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Chi-Joan How, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-566
Record Dates: First submitted 2025-10-16; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: JAK2 Mutation
Keywords: Clonal hematopoiesis; CHIP; JAK2; Myeloproliferative neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ropeginterferon (Experimental)
  Interventions: Drug: Ropeginterferon

INTERVENTIONS:
Drug: Ropeginterferon — Patients will receive Ropeginterferon

SUMMARY:
The goal of this clinical trial is to learn if the drug ropeginterferon alfa-2b can be used safely to treat patients with a JAK2 mutation and high risk features, but do not yet have a myeloproliferative neoplasm. The main questions it aims to answer are:

* Can we enroll 12 patients with JAK2 mutations and high risk features without a myeloproliferative neoplasm on a clinical trial evaluating the drug ropeginterferon?
* Is ropeginterferon safe to use in these patients?

Participants will:

* Receive ropeginterferon as an injection under the skin once every 4 weeks
* Visit the clinic every 1-3 months for checkups and tests

DETAILED DESCRIPTION:
Myeloproliferative neoplasms (MPNs) are driven by dysregulation of the JAK/STAT signaling pathway, most commonly due to the JAK2 V617F mutation. Recent data suggest that JAK2 mutations can arise decades before overt disease, representing an early "precursor" state known as JAK2 clonal hematopoiesis. Individuals with JAK2 clonal hematopoiesis have increased risks of both thrombosis and future MPN development. Early intervention to reduce the malignant clone may therefore improve long-term outcomes.

This is a prospective cohort feasibility study evaluating ropeginterferon alfa-2b in patients with JAK2 V617F clonal hematopoiesis and high-risk features for thrombosis or progression. Participants will receive ropeginterferon by subcutaneous injection every 4 weeks for up to 2 years.

The primary objective is to assess feasibility (enrollment of 12 patients within 2 years) and evaluate the safety and tolerability of ropeginterferon. Secondary objectives include assessing molecular response rates of thrombosis, bleeding, quality of life, and progression to myeloproliferative neoplasm (MPN).

every 6 months through year 2, and again at years 3 and 4 to evaluate durability of response.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years or older
* Evidence of JAK2 V617F clonal hematopoiesis of indeterminate potential, as defined by a JAK2 V617F mutation detected on quantitative PCR. By definition, these patients do NOT have a diagnosis of an MPN, and must have at least one additional high-risk feature.
* Have high-risk clinical/laboratory features, as defined as at least ONE of the following criteria:

  * Patients with a venous or arterial thrombotic event within 1 year of diagnosis of JAK2 clonal hematopoiesis
  * Patients with elevated laboratory parameters above normal limits at screening, but not meeting criteria for an MPN by WHO 2016 criteria. This would include patients with elevated laboratory parameters but an otherwise normal bone marrow biopsy.

    * White blood cell count > 10 K/uL OR
    * Hemoglobin > 16 g/dL in women and > 16.5 g/dL in men; hematocrit >48% for women and >49% for men OR
    * Platelets >400 K/uL
  * Patients with JAK2 VAF >20%
* Willing to have a bone marrow biopsy at study entry to exclude an MPN diagnosis. Screening bone marrow biopsy must not be diagnostic of any overt hematologic malignancy by morphologic assessment and must be consistent with a diagnosis of clonal hematopoiesis as determined by multi-institutional hematopathology review. A historical bone marrow biopsy is allowed if within 3 months of study entry and records and pathology can be obtained. In cases where the bone marrow biopsy results are uncertain, study eligibility should be discussed with the PI. Patients with increased red blood cell parameters or concerning diagnosis for PV should also have an erythropoietin level drawn to assess for a PV diagnosis by WHO 2016 criteria.
* Must have adequate organ function as demonstrated by the following:

  * ALT (SGPT) and/or AST (SGOT) ≤ 2.5x upper limit of normal (ULN), or ≤ 4x ULN (if upon judgment of the treating physician, it is believed to be due to extramedullary hematopoiesis [EMH] related to MF);
  * Direct bilirubin ≤ 1.5 x ULN; or ≤ 2x ULN (if upon judgment of the treating physician, it is believed to be due to extramedullary hematopoiesis [EMH] related to MF);
  * eGFR >60 mL/min
  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * Platelets ≥100,000/mcL
* ECOG performance status (PS) ≤ 3
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* The effects of ropeginterferon on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of ropeginterferon administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Meeting WHO 2016 criteria for a MPN.
* Pregnant or lactating.
* Known history of human immunodeficiency virus (HIV), hepatitis C, or hepatitis B.
* Any active malignancy in the past 2 years, with the exception of non-melanoma skin cancer, or cervical carcinoma in situ or breast carcinoma in situ that has been excised or resected completely and is without evidence of local recurrence or metastasis. Any malignancy treated with curative intent and no evidence for active disease in the last 2 years are eligible.
* Evidence of severe retinopathy or clinically relevant ophthalmologic disorder
* Participation in an investigational drug or device trial within 2 weeks prior to study enrolment
* Documented autoimmune disease at screening or in the medical history which is active and serious
* History of significant and clinically relevant psychiatric illnesses, including prior suicide attempts or risk of suicide on screening
* History of thyroid dysfunction not adequately controlled
* History of major organ transplantation
* History of uncontrolled severe seizure disorder
* Participants who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ropeginterferon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients consented and enrolled within 2 years of study opening | 2 years
  Primary outcome is feasibility, or feasibility of enrolling 12 patients with high-risk JAK2 clonal hematopoiesis onto a clinical trial with ropeginterferon treatment within 2 years of study opening.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 2 years
  Safety and tolerability of ropeginterferon in patients with JAK2 clonal hematopoiesis and high-risk features.

SECONDARY OUTCOMES:
Number of patients with decrease of JAK2 V617F variant allele fraction to undetectable levels if baseline VAF was <10% or decrease of JAK2 V617F VAF by at least 50% if baseline VAF was >10% | 2 years
  Molecular response
Rates of arterial and venous thrombosis | 2 years
Rates of bleeding | 2 years
Patient reported quality of life as measured by the Patient's Impression of Global Change (PGIC) and Patient-Reported Outcomes Measurement Information System 29-item Health Profile (PROMIS-29) | 2 years
Rates of progression to overt MPN | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States